CLINICAL TRIAL: NCT01974336
Title: The Preventative and Therapeutical Effect of Ursodeoxycholic Acid(UDCA) to Parenteral Nutrition-associated Cholestasis in Short Bowel Syndrome
Brief Title: The Preventative and Therapeutical Effect of Ursodeoxycholic Acid(UDCA) to Short Bowel Syndrome Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kong Wencheng, Senior Resident, Jinling Hospital, China
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UDCA-PNAC-SBS
Record Dates: First submitted 2013-10-20; First posted 2013-11-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UDCA+placebo group (Experimental): 15-30mg/kg/d UDCA for 2 months + placebo for 2 months
  Interventions: Drug: ursodeoxycholic acid
- placebo+UDCA (Experimental): placebo for 2 months+15-30mg/kg/d UDCA for 2 months
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Drug: ursodeoxycholic acid

SUMMARY:
The efficacy of UDCA in treating the parenteral nutrition-associated cholestasis(PNAC) has been identified by some studies in children without short bowel syndrome(SBS).Most of the adults who suffering PNAC have SBS. it limits the potential function of UDCA because of the lack of SBS patients and malabsorption of UDCA.Therefore, we design this clinical trial in our center of SBS to approach the preventative and therapeutical effect of UDCA to PNAC in adults with short bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with short bowel syndrome supported by total parenteral nutrition.
* Patients have intestine more than 50cm.
* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Consciousness and ability to cooperate.

Exclusion Criteria:

* Patients have obstruction of biliary tract, infection, autoimmune disease, cancer
* Patients have intestine less than 50cm
* A clinically significant laboratory abnormality or a history of significant cardiac, pulmonary, hepatic, or renal disease
* Female with positive pregnancy
* Allergy to ursodeoxycholic acid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The biochemical indicator of patients' liver function during oral UDCA or placebo | 2 months
  detect the biochemical indicator of patients' liver function(Serum bilirubin, GGT Valley, lactate dehydrogenase, alanine aminotransferase, aspartate aminotransferase) during oral UDCA or placebo

SECONDARY OUTCOMES:
the changs of composition of serum bile acid after oral UDCA or placebo | 2 months
  we test the composition of serum bile acid at the beginning,2 months,4 months(the end) of the trial
The changs of the level of fibroblast growth factor 19(FGF19) in the serum | 4 months
  we test the level of FGF19 in the serum at the beginning,2 months,4months(the end) of the trail.

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Kong, MD, Principal Investigator — Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China